CLINICAL TRIAL: NCT04181307
Title: A Randomized Trial of a BE-EHR Module to Guide the Care of Older Adults With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-01464; 5R33AG057382 (NIH)
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Results first posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard EPIC instantiation (No Intervention): As per standard procedure at NewYorkUniversity Langone Health
- standard EPIC instantiation plus the BE-EHR module. (Experimental): The BE-EHR module includes six components: 1) a tailored advisory for patients over 75 with diabetes, 2) medication refill protocol with information on Choosing Wisely guidelines, 3) pre-population of the medication preference list with metformin, 4) lab result protocol with information on Choosing Wisely guidelines, 5) peer comparisons regarding performance meeting guidelines, and 6) media campaign with information about Choosing Wisely guidelines. The set of nudges is referred to collectively as the BE-EHR module.
  Interventions: Behavioral: BE-EHR module

INTERVENTIONS:
Behavioral: BE-EHR module — The BE-EHR module includes six components: 1) a tailored advisory for patients over 75 with diabetes, 2) medication refill protocol with information on Choosing Wisely guidelines, 3) pre-population of the medication preference list with metformin, 4) lab result protocol with information on Choosing Wisely guidelines, 5) peer comparisons regarding performance meeting guidelines, and 6) media campaign with information about Choosing Wisely guidelines. The set of nudges is referred to collectively as the BE-EHR module.
  Arms: standard EPIC instantiation plus the BE-EHR module.

SUMMARY:
This RCT will test a new electronic health record module to improve guideline-compliant care of older adults with diabetes. The module incorporates effective behavioral economics (BE) principles to improve the degree to which care of older adults is compliant with Choosing Wisely (CW) guidelines; this generally involves less aggressive targets for HbA1c, and reductions of medications other than metformin. The implementation of the module is triggered by patient scheduling and medication prescribing in EPIC. The BE principles include suggesting alternatives to medications, requiring justification, setting of appropriate default order sets, and incorporation of anchoring and checklists to guide behavior.

ELIGIBILITY:
Inclusion Criteria:

* Patient at NYULH primary care or endocrinology practice
* Practices that have patients aged 75 or older
* Practices that have a diagnosis of diabetes in the EHR chart

Exclusion Criteria:

• Under age 75

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 7630 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Troxel, ScD, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to andrea.troxel@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Viswanadham RVN, Belli HM, Martinez TR, Wong C, Blecker S, Troxel AB, Mann DM. When Nudges Don't Budge: A Mixed Methods Study of Why EHR-Based Deprescribing Nudges Failed to Change Provider Behavior. Res Sq [Preprint]. 2025 Sep 23:rs.3.rs-7466262. doi: 10.21203/rs.3.rs-7466262/v1. PMID 41041570
- [Derived] Belli HM, Troxel AB, Blecker SB, Anderman J, Wong C, Martinez TR, Mann DM. A Behavioral Economics-Electronic Health Record Module to Promote Appropriate Diabetes Management in Older Adults: Protocol for a Pragmatic Cluster Randomized Controlled Trial. JMIR Res Protoc. 2021 Oct 27;10(10):e28723. doi: 10.2196/28723. PMID 34704959

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard EPIC Instantiation | Standard EPIC Instantiation Plus the BE-EHR Module.
Started | 2986 | 4644
Assessed at Baseline | 1342 | 2086
Assessed at 18 Months | 1644 | 2558
Completed | 1342 | 2086
Not Completed | 1644 | 2558

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard EPIC Instantiation | Standard EPIC Instantiation Plus the BE-EHR Module. | Total
Number analyzed (Participants) | 1342 | 2086 | 3428
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.8 (4.5) | 81.4 (4.6) | 81.6 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 776 | 1096 | 1872
  Male | 566 | 990 | 1556
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 240 | 189 | 429
  Not Hispanic or Latino | 955 | 1624 | 2579
  Unknown or Not Reported | 147 | 273 | 420
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 3 | 9
  Asian | 42 | 71 | 113
  Native Hawaiian or Other Pacific Islander | 6 | 4 | 10
  Black or African American | 112 | 282 | 394
  White | 948 | 1501 | 2449
  More than one race | 0 | 6 | 6
  Unknown or Not Reported | 228 | 219 | 447
Region of Enrollment [Number; unit: participants]
  United States | 1342 | 2086 | 3428

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are CW-Compliant and CW-Noncompliant
Description: In order to evaluate Choosing Wisely (CW) compliance status, the BE-EHR algorithm will capture information on demographics, diagnoses in the patient's problem list, prescription history, and relevant lab results (i.e. allergies and blood glucose (HbA1c)) The study team members will not collect this information directly; data will be collected in NYULH's EHR system, EPIC, and an EPIC Reporting analyst will extract the relevant parameters from the EHR into a report. The study team members only receive the ultimate determination from the algorithm that the patient is either CW-compliant or CW-noncompliant.
Time Frame: Month 18
Measure: Count of Participants; unit: Participants
Arm/Group | Standard EPIC Instantiation | Standard EPIC Instantiation Plus the BE-EHR Module.
Number analyzed (Participants) | 1644 | 2558
Participants
  CW-Compliant | 412 | 704
  CW-Noncompliant | 1232 | 1854

2. Secondary Outcome: Number of Total Prescription Encounters
Description: The Refill Protocol nudge activates in Epic any time a medication refill for either Metformin or a non-Metformin diabetes medication is generated for a patient over 75
Time Frame: Month 18
Measure: Number; unit: Prescription Encounters
Arm/Group | Standard EPIC Instantiation | Standard EPIC Instantiation Plus the BE-EHR Module.
Number analyzed (Participants) | 1644 | 2558
Prescription Encounters | 0 | 2056

ADVERSE EVENTS:
Time Frame: 18 months
Description: Study team monitors adverse events via patient's Electronic Health Record.
Arm/Group | Standard EPIC Instantiation | Standard EPIC Instantiation Plus the BE-EHR Module.
All-Cause Mortality (participants affected / at risk) | 18/1644 | 21/2558
Serious Adverse Events (participants affected / at risk) | 0/1644 | 0/2558
Other Adverse Events (participants affected / at risk) | 0/1644 | 0/2558

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT04181307/Prot_SAP_000.pdf